CLINICAL TRIAL: NCT01986608
Title: A Single Center Open-label, Randomized, Single-dose, 3-way Crossover Study to Compare the Safety, Tolerability, and Pharmacokinetics of Lacosamide Administered as Oral Tablet or Intravenous Infusion in Healthy Japanese Subjects
Brief Title: Bioavailability/Bioequivalence Study Between Lacosamide Tablet and Solution for Infusion in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: EP0036; 2012-003084-21 (EudraCT Number)
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Healthy Volunteers
Keywords: Lacosamide; Vimpat; Bioequivalence; Bioavailability; Japanese
MeSH Terms: interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lacosamide 30-minute iv (Experimental): A 30-minute intravenous constant infusion of Lacosamide (LCM) 200 mg (200 mg/20 mL single-use vial).
  Interventions: Drug: Lacosamide infusion
- Lacosamide 60-minute iv (Experimental): 60-minute intravenous constant infusion of Lacosamide (LCM) 200 mg (200 mg/20 mL single-use vial).
  Interventions: Drug: Lacosamide infusion
- Lacosamide oral tablet (Experimental): Oral administration of Lacosamide (LCM) 200 mg (2 x 100 mg film-coated tablet) with 200 mL of water.
  Interventions: Drug: Lacosamide oral

INTERVENTIONS:
Drug: Lacosamide infusion — Strength: 10 mg/mL for infusion
  Form: solution for infusion
  Dosage: 200 mg, single dose
  Duration: 30-minute infusion or 60-minute infusion
  Other Names: Vimpat
  Arms: Lacosamide 30-minute iv; Lacosamide 60-minute iv
Drug: Lacosamide oral — Strength: 200 mg
  Form: film-coated tablet
  Dosage: 200 mg, single dose
  Duration: single oral intake
  Other Names: Vimpat
  Arms: Lacosamide oral tablet

SUMMARY:
This study will be conducted to compare the pharmacokinetics of Lacosamide (LCM) following a single 30-minute or 60-minute iv infusion of LCM 200 mg with those following a single oral dose of LCM 200 mg in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male and female volunteers with the age between 20 and 55 years old

Exclusion Criteria:

* Subject has participated or is participating in any other clinical studies of investigational drug or another investigational medical product within the last 3 months
* Subject has a history (within 6 months) before screening visit of chronic alcohol and/or drug abuse and/or has smoked and/or has a history or presence of cardiovascular, respiratory, hepatic, renal, GI, endocrinological, or neurological disorders
* Subject has a history of suicide attempt or current active suicidal ideation
* Subject has experienced a myocardial infarction and/or made a blood donation or any other blood loss more than 400 ml in the last 3 months
* Subject is pregnant or nursing
* Subject is not healthy (eg, taking any drug treatments, having any medical or emotional/psychological problems, a drug/alcohol abuse, having abnormal safety parameters and/or was positive for HIV, HBsAg, HCV)
* Subject has an excessive use of alcohol or/and cigarettes and/or caffeine and/or abnormal diet and/or has taken grapefruit or grapefruit drink within 7 days before intake of Investigational Medicinal Product (IMP)
* Subject has a clinically significant abnormality in the 12-lead Electrocardiogram (ECG)
* Subject is having clinically relevant drug hypersensitivity to any components of the investigational medicinal product

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of Lacosamide (Cmax) after oral and intravenous administration of Lacosamide | Pharmacokinetic samples will be taken at predose/preinfusion, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours postdose (start of infusion)
Area under the plasma concentration-time curve from zero up to the last analytically quantifiable concentration of Lacosamide (AUC 0-t) after oral and intravenous administration of Lacosamide | Pharmacokinetic samples will be taken at predose/preinfusion, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours postdose (start of infusion)

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from zero up to infinity (AUC) after oral and intravenous administration of Lacosamide | Pharmacokinetic samples will be taken at predose/preinfusion, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours postdose (start of infusion)
Time to reach a maximum plasma concentration (tmax) after oral and intravenous administration of Lacosamide | Pharmacokinetic samples will be taken at predose/preinfusion, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours postdose (start of infusion)
Mean residence time (MRT) after oral and intravenous administration of Lacosamide | Pharmacokinetic samples will be taken at predose/preinfusion, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours postdose (start of infusion)
Rate constant of elimination (λz) after oral and intravenous administration of Lacosamide | Pharmacokinetic samples will be taken at predose/preinfusion, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours postdose (start of infusion)
Terminal half-life (t1/2) after oral and intravenous administration of Lacosamide | Pharmacokinetic samples will be taken at predose/preinfusion, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours postdose (start of infusion)
Apparent total body clearance (CL/F) after oral administration of Lacosamide | Pharmacokinetic samples will be taken at predose/preinfusion, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours postdose (start of infusion)
Total body clearance (CL) after intravenous administration of Lacosamide | Pharmacokinetic samples will be taken at predose/preinfusion, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours postdose (start of infusion)
Apparent volume of distribution (Vz/F) after oral administration of Lacosamide | Pharmacokinetic samples will be taken at predose/preinfusion, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours postdose (start of infusion)
Volume of distribution (Vz) after intravenous administration of Lacosamide | Pharmacokinetic samples will be taken at predose/preinfusion, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, and 72 hours postdose (start of infusion)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- 001, Harrow, Middlesex, United Kingdom